CLINICAL TRIAL: NCT04724096
Title: Evaluation of Oxygen Enhanced Magnetic Resonance Imaging for Identification of Hypoxia Induced Resistant Tumours in Patients With Head and Neck Cancer
Brief Title: Evaluation of OE-MRI in Patients With H&N Cancer
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20MP001
Record Dates: First submitted 2021-01-21; First posted 2021-01-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Oxygen enhanced MRI
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-patient volunteers: 5 non-patient volunteers for testing of protocol to allow for the ascertaining of good quality data prior to the scanning of patients.
  Interventions: Diagnostic Test: Oxygen Enhanced MRI scan
- Patients: 50 patients to be scanned with the oxygen enhanced MRI scan protocol prior to definitive curative intent therapy.
  Interventions: Diagnostic Test: Oxygen Enhanced MRI scan

INTERVENTIONS:
Diagnostic Test: Oxygen Enhanced MRI scan — Dynamic MRI scanning switching from breathing room air to high concentration oxygen part way through the scan.

SUMMARY:
Assessment of the use of oxygen enhanced MRI scanning in a cohort of patients with head and neck squamous cell carcinomas to identify areas of hypoxia with tumours and relate this to treatment outcomes.

DETAILED DESCRIPTION:
Oxygen-enhanced MRI (OE-MRI) is a technique being actively investigated for imaging hypoxia within cancer tissues. Preliminary clinical data demonstrates the feasibility of using this methodology to study patients with head and neck squamous cell carcinoma (HNSCC). The investigators wish to investigate using this methodology to identify hypoxic subvolumes within HNSCC that may have greater resistance to standard radiotherapy treatment and investigate the association of such hypoxic regions with treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Non-patient Volunteer Inclusion Criteria:

* Age 18 years and above
* Signed written informed consent

Patient Inclusion Criteria:

* Histologically proven or strong clinical suspicion of squamous cell carcinoma of the head and neck
* Suitable for undergoing radical radiotherapy or chemoradiotherapy according to local protocols within the head and neck Cancer MDT
* Age 18 years and above
* Adequate physical fitness (WHO performance status 0 to 2)
* Signed written informed consent

Exclusion Criteria:

Non-patient Volunteer Exclusion Criteria:

* Contraindications to MRI scans as identified following completion of the Nottingham University Hospitals NHS Trust (NUH) standard MR safety screening protocol
* Severe Chronic Obstructive Pulmonary Disease (COPD) who are at risk of type 2 respiratory failure or require supplemental oxygen
* Volunteers who are pregnant as identified through the NUH standard MR safety screening protocol

Patient Exclusion Criteria:

* Poor physical fitness (WHO performance status greater than 2)
* Contraindications to MRI scans as identified following completion of the NUH standard MR safety screening protocol
* Severe Chronic Obstructive Pulmonary Disease (COPD) who are at risk of type 2 respiratory failure or require supplemental oxygen
* Patients who are pregnant or breast-feeding (due to IV contrast use in the routine clinical scan) as identified through the NUH standard MR safety screening protocol

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 5 non-patient volunteers. 50 patients from Nottingham University Hospitals NHS Trust, UK.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with areas detected within tumours of the head and neck area that have measurable hypoxia using OE-MRI technique. | 2 years
  Feasibility of OE-MRI scans to detect hypoxic areas within tumours in patients with head and neck squamous cell carcinomas
Association with treatment failure | 2 years
  Test predictive value of OE-MRI to identify patients with the highest risk of treatment failure and provide data to allow a power calculation for a larger future trial of the predictive power of OE-MRI for treatment outcomes in head and neck cancer treated with radiotherapy.

SECONDARY OUTCOMES:
Tumour perfusion | 2 years
  Assessment of routinely used diagnostic MRI images to identify non-perfused parts of tumours in combination with oxygen maps

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Panek, PhD, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Queens Medical Centre, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McCabe A, Martin S, Rowe S, Shah J, Morgan PS, Borys D, Panek R. Oxygen-enhanced MRI assessment of tumour hypoxia in head and neck cancer is feasible and well tolerated in the clinical setting. Eur Radiol Exp. 2024 Mar 6;8(1):27. doi: 10.1186/s41747-024-00429-1. PMID 38443722